CLINICAL TRIAL: NCT00358371
Title: A Mono-center, Open, Randomized, Three-way, Twelve-sequence, Cross-over Study to Determine the Extent of Absorption (Absolute Bioavailability), Rate of Absorption and to Further Characterize Distribution and Elimination Characteristics of a Commercial 250 mg and a 500 mg Capsule of Flucloxacillin Each Given as a Single Oral Dose vs. One 250 or 500 mg Intravenous Dose to 24 Healthy Male and/or Female Subjects in the Fasting State
Brief Title: Bioavailability Of Flucloxacillin Capsules (250 mg and 500 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 103811
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Infections, Bacterial
Keywords: bioavailability flucloxacillin
MeSH Terms: conditions — Bacterial Infections | interventions — Floxacillin

ARMS (2):
- Subjects receiving flucloxacillin 250 mg (Experimental): Subjects will be randomized to receive single oral dose of 250 mg flucloxacillin capsule and 250 mg Intravenous dose
  Interventions: Drug: flucloxacillin 250 mg
- Subjects receiving flucloxacillin 500 mg (Experimental): Subjects will be randomized to receive single oral dose of 500 mg flucloxacillin capsule and 500 mg Intravenous dose
  Interventions: Drug: flucloxacillin 500 mg

INTERVENTIONS:
Drug: flucloxacillin 250 mg — Subjects will be randomized to receive single oral dose of 250 mg flucloxacillin capsule and 250 mg Intravenous dose
  Other Names: flucloxacillin
  Arms: Subjects receiving flucloxacillin 250 mg
Drug: flucloxacillin 500 mg — Subjects will be randomized to receive single oral dose of 500 mg flucloxacillin capsule and 500 mg Intravenous dose
  Arms: Subjects receiving flucloxacillin 500 mg

SUMMARY:
Primary objective:To study the absolute bioavailability, distribution and elimination parameters of flucloxacillin from two oral formulations of flucloxacillin in healthy male and/or female subjects.

DETAILED DESCRIPTION:
A mono-center, open, randomized, three-way, twelve-sequence, cross-over study to determine the extent of absorption (absolute bioavailability), rate of absorption and to further characterize distribution and elimination characteristics of a commercial 250 mg and a 500 mg capsule of flucloxacillin each given as a single oral dose vs. one 250 or 500 mg intravenous dose to 24 healthy male and/or female subjects in the fasting state

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* Caucasians,
* Body Mass Index (BMI) between 19 and 27 kg/m 2;
* physically and mentally healthy as judged by means of a medical and standard lab examination;
* non-smokers,
* ex-smokers or moderate smoker.

Exclusion criteria:

* medical history,
* vital signs,
* physical examination,laboratory tests (blood and/or urine) with evidence of clinically significant conditions;
* 12-lead electrocardiogram (ECG) with clinically significant abnormality;acute infection within 2 weeks preceding 1st study drug administration;any medication on a regular basis (exception females: oral contraceptives) and/or tricyclic antidepressants, antacids, histamine H2-receptor antagonists, antibiotics,
* non steroid anti-inflammatory drugs or anticoagulants within 8 weeks before the 1st study drug administration and/or no agreement to take any of those drugs including Over-the-counter (OTC) drugs until the end of the follow- up examination;
* no agreement not to take any medication,including OTC medicine, antacids, or analgesics within 2 weeks before 1st drug administration until the end of the follow-up examination;special diet or loss of > 5 kg within last month from a weight reduction diet; regularly consume of large quantities of alcohol (> 20g/day) and/or beverages containing methylxanthines e.g. caffeine (> 0.5L/day altogether);
* no agreement not to consume: - any beverages or foods containing alcohol 48 h prior to 1st study drug administration until end of the follow-up examination;
* any grapefruit products 7 days prior 1st study drug administration until end of the follow-up examination,
* any beverages or foods containing methylxanthines as well as fruit-juices and any foods containing poppy seed 48 h before 1st drug administration of either study period until last blood sample of the respective study period was collected,
* not to consume chewing during confinement;
* history of: - allergy to flucloxacillin,
* B-lactams and/or related drugs,
* known hypersensitivity against the inactive ingredients of the study medication,
* hypersensitivity to multiple drugs,
* allergic diseases,
* acute hay fever,
* previous history of flucloxacillin-associated jaundice/hepatic dysfunction,
* alcohol or drug abuse,
* epilepsy or other seizure,
* psychiatric illness, e.g. latent or manifest depression schizophrenia, or neurosis,
* respiratory diseases,
* surgery of the gastrointestinal tract (except appendectomy),
* kidney diseases,
* bleeding/coagulation disorder or severe anaemia,
* glucose-6-phosphate dehydrogenase deficiency and/or chronic treatment or chronic pathology;
* metabolic disease;
* evidence for disorder in the metabolism of pharmaceuticals or other foreign compounds; cardiovascular diseases e.g. hypertension, hypotension or bradycardia;
* associated disease that would interfere with the clinical course of the trial;
* major illness during 3 month before commencement of the screening period,
* gastrointestinal diseases;
* reported or positive results from test of drugs of abuse (amphetamines, opiates, barbiturate, methadone, cannabinoids, cocaine, benzodiazepines);
* Positive test for: alcohol, Hepatitis-B-antigen or Hepatitis-C-antibody, HIV-antibody;blood donor or blood loss including plasmapheresis within the last 3 months before the 1st study drug administration;
* intake of depot injectable solutions (including study medication) within 6 month before 1st study administration;
* intake of enzyme-inducing and/or organotoxic drugs within 4 weeks before 1st study drug administration;for females only: positive results from pregnancy tests;does not use or not agree to use adequate contraceptive methods during the study;
* lactating woman.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01-06 (Actual); Primary Completion 2005-02-08 (Actual); Study Completion 2005-02-08 (Actual)

PRIMARY OUTCOMES:
Absolute (Abs.) bioavailability, max. plasma conc., concentration-time curve (AUC) from 0 hto the last quantifiable conc., AUC from 0 h to infinity), timepoint of max. plasma conc., Halflife of drug elimination during the terminal phase | Up to 60 Days

SECONDARY OUTCOMES:
Elimination rate constant, total Clearance, Volume of distribution at steady state, Volume of distribution during the terminal phase, residual area | Up to 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- See also: Results for study 103811 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/103811?search=study&search_terms=103811#rs